CLINICAL TRIAL: NCT04321369
Title: Impact of Swab Site and Sample Collector on Testing Sensitivity for COVID-19 Virus in Symptomatic Individuals
Status: Completed | Type: Observational
Sponsor: UnitedHealth Group (Industry)
Collaborators: Quest Diagnostics-Nichols Insitute (Industry); Bill and Melinda Gates Foundation (Other)
Responsible Party: Sponsor
Other Study IDs: 20-001
Record Dates: First submitted 2020-03-23; First posted 2020-03-25 (Actual); Last update posted 2022-05-04 (Actual); Status verified 2022-04

CONDITIONS: Infections, Respiratory; Fever; Cough
MeSH Terms: conditions — Respiratory Tract Infections; Fever; Cough

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Biospecimen Retention: None Retained — Four nasal swabs will be collected on each participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Testing Sensitivity for SARS-CoV-2 Virus in Symptomatic Individuals — This is an operational project. Patients will collect a sample from the tongue, nasal cavity and MT and then clinicians will collect a NP sample from the nostril corresponding to each participant's dominant hand.

SUMMARY:
Operational project to compare clinician collected nasopharyngeal (NP) samples to patient-obtained tongue, nasal and mid-turbinate (MT) samples in the detection of SARS-CoV-2 in an outpatient clinic setting

DETAILED DESCRIPTION:
This work will serve both the Everett Clinic and broader UnitedHealth Group patient populations as well as advance the public health emergency (PHE) response to the community spread of SARS-CoV-2 virus, especially as the number of cases and deaths continues to rise in many geographies. Leveraging our presence in the Seattle/Puget Sound area with Everett Clinic, we intend to develop a model that can screen a large number of patients at varying levels of risk and manifestation of clinical symptoms while conserving personal protective equipment (PPE) and decreasing transmission risk to health care workers. This will also serve to support the enterprise and public health response. Towards this goal, we must first assess the equivalence between clinician-collected nasopharyngeal (NP) samples to patient-collected tongue, nasal, and mid-turbinate (MT) samples to detect SARS-CoV-2 across a broad cross-section of the population.

ELIGIBILITY:
Inclusion Criteria:

* Able to consent and agree to participate in the project after discussing the project
* Coming to The Everett Clinic during the operational project duration
* Evidence of upper respiratory symptoms suggesting higher risk of testing positive for SARS-CoV-2 virus.

Exclusion Criteria:

* Not able to demonstrate understanding of the study
* Not willing to commit to having all four samples collected
* Medical history evidencing any of the following

  * Active nosebleed in the past 24 hours
  * Nasal surgery in the past two weeks
  * Chemotherapy treatment with low platelet and low white blood cell counts
  * Acute facial trauma

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients presenting symptoms indicative of an upper respiratory infection visiting one of the five Everett Clinic sites of during the study duration while the operational project is occurring are eligible to participate in the project.
Sampling Method: Non-Probability Sample
Enrollment: 530 (Actual)
Dates: Start 2020-03-09 (Actual); Primary Completion 2020-03-23 (Actual); Study Completion 2020-03-23 (Actual)

PRIMARY OUTCOMES:
Accuracy of patient administered tests | 2 weeks
  compare clinician collected nasopharyngeal (NP) samples to patient-obtained tongue, nasal and mid-turbinate (MT) samples in the detection of SARS-CoV-2 in an outpatient clinic setting

CONTACTS AND LOCATIONS:
Overall Officials: Ethan Berke, MD, Principal Investigator — UnitedHealth Group
Locations (1):
- Everett Clinic, Seattle, Washington, United States

IPD SHARING:
Plan to Share IPD: Yes
All patients who participate in this operational pilot will have standard COVID-19 screening information entered into their electronic medical record. The collection locations and source of collection (medical personnel versus patient) will need to be clearly distinguished for the purposes of this project. Data resulting from analysis of the samples will also be stored in the electronic medical record and any positive results will be reported accordingly to public health officials as required. The data collected due to this operational effort will be extracted from the medical record and stored for additional research analysis to demonstrate equivalence between location in the nose for the collection of the sample and similarity between sample collected by medical personnel and samples collected by the patient. Data will be shared between the participating clinics, UHG and collaborating partners performing the analysis of the samples and returning results.
Supporting Information: Study Protocol
Time Frame: March 2020 - June 2020
Access Criteria: . Data will be shared between the participating clinics, UHG and collaborating partners performing the analysis of the samples and returning results as outlined in data sharing agreements.

REFERENCES:
- [Result] Coronavirus Disease 2019 (COVID-19) in the US. Centers for Disease Control and Prevention, accessed March 13, 2020. https://www.cdc.gov/coronavirus/2019-ncov/cases-in-us.html
- [Result] Personal communication per Dr. Scott Lindquist, MD State of Washington Epidemiologist (March 2020
- [Result] Anderson RM, Heesterbeek H, Klinkenberg D, Hollingsworth TD. How will country-based mitigation measures influence the course of the COVID-19 epidemic? Lancet. 2020 Mar 21;395(10228):931-934. doi: 10.1016/S0140-6736(20)30567-5. Epub 2020 Mar 9. No abstract available. PMID 32164834
- [Result] Frazee BW, Rodriguez-Hoces de la Guardia A, Alter H, Chen CG, Fuentes EL, Holzer AK, Lolas M, Mitra D, Vohra J, Dekker CL. Accuracy and Discomfort of Different Types of Intranasal Specimen Collection Methods for Molecular Influenza Testing in Emergency Department Patients. Ann Emerg Med. 2018 Apr;71(4):509-517.e1. doi: 10.1016/j.annemergmed.2017.09.010. Epub 2017 Nov 24. PMID 29174837

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-03-13): https://cdn.clinicaltrials.gov/large-docs/69/NCT04321369/Prot_SAP_000.pdf